CLINICAL TRIAL: NCT00417664
Title: ICU Delirium: Can Dexmedetomidine Reduce Its Incidence?
Brief Title: Is Dexmedetomidine Associated With a Lower Incidence of Postoperative Delirium When Compared to Propofol or Midazolam in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 77815
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Delirium
Keywords: cardiac surgery; valvular surgery; delirium; postoperative delirium; cognitive dysfunction; altered mental status
MeSH Terms: conditions — Delirium; Emergence Delirium; Cognitive Dysfunction | interventions — Dexmedetomidine; Propofol; Midazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Propofol
  Interventions: Drug: Propofol
- Midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine administered as part of anesthesia in cardiac surgery patients
  Other Names: Precedex
  Groups: Dexmedetomidine
Drug: Propofol — Propofol administered as part of anesthesia in cardiac surgery patients
  Groups: Propofol
Drug: Midazolam — Midazolam administered as part of anesthesia in cardiac surgery patients
  Groups: Midazolam

SUMMARY:
The purpose of this chart review study is to determine whether the use of dexmedetomidine, a selective α2-adrenergic receptor agonist with sedative, analgesic, and antinociceptive properties, would be associated with a lower incidence of delirium when compared to propofol and midazolam. We hypothesize that sedation with dexmedetomidine following cardiac surgery with CPB will be associated with a lower incidence of postoperative delirium.

DETAILED DESCRIPTION:
Delirium is the most common psychiatric syndrome found in the general hospital setting. Between 32 - 80% of cardiac surgery patients may experience post-operative delirium. Because failure to recognize delirium leads to increased morbidity and mortality and prolonged hospital stays, there are compelling clinical and financial reasons to improve the identification and treatment of delirium. Dexmedetomidine, a selective alpha2-adrenergic receptor agonist, may be an alternative to current postoperative sedation when it comes to lowering the incidence of delirium.

Comparisons: The use of postoperative (at sternal closure) dexmedetomidine will be compared to current standards of care propofol and midazolam for postoperative sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a coronary artery disease, cardiac valve disease, or vascular problems requiring elective surgical intervention
2. Age older than 18 years of age, less than 90 years of age
3. Fluency in English, and willingness to participate in the study
4. No history of recent (< 3 months) of alcohol or drug abuse
5. No pre-operative evidence of heart block
6. No history of dementia, schizophrenia, or post-traumatic stress disorder

Exclusion Criteria:

1. A preexisting diagnoses of dementia, schizophrenia, active or recent alcohol or drug abuse/dependence; post-traumatic stress disorder; acute intoxication (i.e., positive urine drug and/or alcohol test at the time of initial evaluation or upon hospitalization for surgery)
2. Age younger than 18, or older than 89 years of age
3. Inability to understand enough English to complete required diagnostic testing
4. Unwillingness to participate in the study
5. Inability of subject or surrogate to consent.
6. Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2002-04; Primary Completion 2004-01 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Postoperative Delirium (DSM-IV criteria)

SECONDARY OUTCOMES:
Length of Stay (hospital and ICU), use of as needed medications

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Maldonado, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States